CLINICAL TRIAL: NCT07361458
Title: Modex, a Cloud-based, Centralized Health Economic Model Marketplace to Reduce Costs and Enhance Equity in Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arnold Consultancy & Technology, LLC (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Renee JG Arnold, PharmD, President and CEO, Arnold Consultancy & Technology, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R43CA297808-01 (NIH); 1R43CA297808-01 (NIH)
Record Dates: First submitted 2025-12-06; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: oncology; model; health economics; open source model; open source; prototype; wireframes
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Advisory Panelist participants will be randomly assigned to interact with wireframes of the prototype and then several models according to key use cases (e.g. model publishing, model searching, user registration, user profile updating, payments, etc.), and then provide answers to the System Usability Scale questions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advisory Panelist participa will evaluate wireframes and a working prototype of the HModEx® website. (Other): This is a single-arm study that will build and evaluate (via usability testing) an open source health economic model platform prototype using a 9-member expert advisory panel of health economist participants from the US and Europe.
  Interventions: Other: open source health economic models

INTERVENTIONS:
Other: open source health economic models — open source health economic models

SUMMARY:
The investigators intend to create and test an interactive prototype of an online health economic model platform, ModEx™ (renamed HModEx®), to house oncology models. The primary objective is to create the HModEx® health economic model platform. The secondary objective is to conduct usability testing of search, quality and collaboration on the HModEx® prototype for 20 oncology health economic models with expert advisory panel participants.

DETAILED DESCRIPTION:
Primary Endpoint: Iteratively unit test 4 tasks (A) Revise model platform and back end, (B) Refine the model taxonomy/characterization (i.e., ontology) and search module, (C) Revamp submission module, and (D) Implement paid modules) individually to ascertain 100% pass of common functionality (e.g., searching, uploading, and evaluating models) in the system back end and then iteratively perform integration testing via the front-end user interface until 100% pass using the System Usability Scale (as below). The System Usability Scale yields a single number representing a composite measure of the overall usability of the system being studied. To calculate the System Usability Scale score, first sum the score contributions from each item. Each item's score contribution will range from 0 to 4. For items 1,3,5,7, and 9 the score contribution is the scale position minus 1. For items 2,4,6,8 and 10, the contribution is 5 minus the scale position. Multiply the sum of the scores by 2.5 to obtain the overall value of System Usability Score; scores range from 0 to 100, with higher numbers being better.

Secondary Endpoints: Measure the success of Aim 2 by (1) completion of 80% of tasks in usability testing with scores of ≥68 on the System Usability Scale, a validated questionnaire, and (2) satisfaction with the site. Testing will focus on user interaction with the system, emphasizing effectiveness, efficiency, engagingness, error tolerance, and ease of learning. Specifically, the investigators will assess the ability of the project team and Advisory Panel member participants to log into the platform, configure and manage their modeling projects, and annotate or categorize them in accordance with an ontological index. The investigators will assign participants to interact with at least 2 randomly selected models and associated data files, iterating on this milestone until the investigators achieve 100% success.

ELIGIBILITY:
Inclusion Criteria:

* Expert Advisory Panel member

Exclusion Criteria:

* Non-English-speaker

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Alpha testing of wireframe usability | 2 months
  Iteratively unit test 4 tasks (A) Revise model platform and back end, (B) Refine the model taxonomy/characterization (i.e., ontology) and search module, (C) Revamp submission module, and (D) Implement paid modules) individually to ascertain 100% pass of common functionality (e.g., searching, uploading, and evaluating models) in the system back end and then iteratively perform integration testing via the front-end user interface until 100% pass using the System Usability Scale. The overall value of the System Usability Score ranges from 0 to 100. The higher the score on the System Usability Scale, the better.

SECONDARY OUTCOMES:
Beta testing of prototype usability | 4 months
  Measure the success of Aim 2 by (1) completion of 80% of tasks in usability testing with scores of ≥68 on the System Usability Scale, a validated questionnaire, and (2) satisfaction with the site. Testing will focus on user interaction with the system, emphasizing effectiveness, efficiency, engagingness, error tolerance, and ease of learning. Specifically, the investigators will assess the ability of the project team and Advisory Panel member participants to log into the platform, configure and manage their modeling projects, and annotate or categorize them in accordance with an ontological index. The investigators will assign panelist participants to interact with at least 2 randomly selected models and associated data files, iterating on this milestone until the investigators achieve 100% success. The overall value of the System Usability Score ranges from 0 to 100. The higher the score on the System Usability Scale, the better.

CONTACTS AND LOCATIONS:
Overall Officials: Renee JG Arnold, PharmD, Principal Investigator — Arnold Consultancy & Technology, LLC
Locations (1):
- Arnold Consultancy & Technology, LLC, Miami Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Actually, this will be aggregated System Usability Score data that will be shared with other researchers and the backgrounds, but not the individual identities, of the participants will be disclosed in presentations and publications.

DOCUMENTS (1):
  • Study Protocol (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT07361458/Prot_000.pdf